CLINICAL TRIAL: NCT02595164
Title: Common Decision Making Deficits in Suicidal Behaviors and Eating Disorders
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Schneider Children's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SHEBA-15-2191-EGA-CTIL
Record Dates: First submitted 2015-07-19; First posted 2015-11-03 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-11

CONDITIONS: Anorexia Nervosa; Bulimia Nervosa; Suicide; Parasuicide; Self-Injurious Behavior; Impulsive Behavior
MeSH Terms: conditions — Anorexia Nervosa; Bulimia Nervosa; Suicide; Suicide, Attempted; Self-Injurious Behavior; Impulsive Behavior

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Impulsive subjects: Subjects exhibiting impulsive symptoms Behavioral Task
- Non-impulsive subjects: Subjects which do not exhibit impulsive symptoms Behavioral Task

SUMMARY:
The role of impulsivity and its contribution to suicidal behavior seems intuitively clear. Empirical results have proved the existence of a relationship between the two yet many questions are left unanswered, especially what differentiates suicide ideators from attempters.. Obsessive thinking patterns are thought processes which share a repetitive behavior domain and are exerted by an inner voice. 3 types of obsessive thinking patterns are self destructive thoughts, ruminations and overvalued ideas. Impulsivity and obsessive thinking patterns are presumed to have a common mechanism of behaviors which are resulted from basal ganglia dysregulation and thus effect inhibition. Novel research in the field of decision making could help to learn more about behavioral patterns associated with self harm behavior and suicide. Eating Disorders involve suicidal and self harm behavior, which both feature impulsivity and obsessive thinking patterns. The investigators study proposes a 3-step theoretical model which asserts there is a connection between impulsivity, obsessive thinking and poor decision making, all effecting self harm behavior. Contemporary research has not been able to fully understand the nature of impulsivity and its effect on self harm behavior, including eating disorders symptoms, nor addressed the impact of obsessive thinking patterns on the latter. 100 female participants with Eating Disorders and suicidal behavior will be recruited for the proposed research. Subjects will be given self-report questionnaires and computerized behavioral tasks. A one way ANOVA of two eating disorder subgroups, impulsive and non impulsive, will be conducted, following a hierarchical multiple regression with self harm behavior being the dependent variable.

DETAILED DESCRIPTION:
Aim of Study impulsivity and its relation to different self harm behaviors, specifically suicidal attempts, is an ongoing field of study which has already been widely discussed. Yet to this date, the relationship remains unclear and somewhat confusing. Possible explanations for this might be due to the fact that impulsivity is an ill-defined concept leading to numerous definitions used by different studies and the fact that it has a trait and state aspect to it. Clinical experience and theory leads to the assumption that impulsivity plays a very important role in suicide. Novel research in the field of decision making could possibly lead to a breakthrough in improving assessment and prevention of suicide attempts and learning more of this complex relationship.

The study of obsessive thinking patterns and their contribution to suicide is less prominent. In spite of the lack of magnitude in research, when looking at underlying mechanisms it is noticeable that both impulsivity and obsessive thinking share common factors and are congruent in many ways. Determining more about the nature of different obsessive thinking patterns such as self destructive thoughts, rumination and over-valued ideas manifested by an inner voice is crucial from two points of view: on one hand learning more about the relation between the different patterns, and their mutual and independent effect on self harm behavior. On the other hand, observing them as complementing factors to impulsivity which may lead to a better understanding of the latter. Studying the interaction between trait impulsivity and different obsessive thinking patterns could lead to a better understanding of the theoretical gap discussed in the literature review between suicidal ideators and attempters.

Literature has proven that observing behavioral patterns in decision making tasks could serve as a better predictor to self harm and suicidal behavior, compared to solely relying on self report. The investigators intention is to try and find correlations between the personality dimensions of impulsivity and obsessive thinking and specific behavioral patterns indicating suicidal and self harm behavior. Understanding more on impulsive and obsessive thinking patterns and their effect on self harm behaviors in "real life" situations can raise the ecological validity and aid in exporting research conclusions to a clinical setting.

The investigators research will recruit a population which is known to feature both impulsivity and obsessive thinking patterns, such as in Eating Disorders, where their co-existence has been proven empirically yet the nature of the interaction is not fully understood. Eating disorder individuals are also at higher risk of attempting suicide and exhibiting self harm behaviors in general compared to a non clinical population, making it a relevant group to the proposed study.

The investigators propose that impulsive behavior and obsessive thinking patterns have a negative effect on performance in decision making situations. When there is a tendency to make bad decisions the risk of executing different forms of self harm rises, including suicidal behavior and eating disorders.

Method:

Participants The investigators will recruit 100 participants from a sample of female patients, diagnosed with Eating Disorders and suicidal behavior, admitted to mental health departments in general and psychiatric hospitals. Diagnosis will be made by the hospital staff. After receiving approval from the medical staff participants will be interviewed, handed questionnaires and computerized tasks.

Procedure Research will consist of two parts: at first investigators will conduct a preliminary research on 20 subjects which is intended to decrease questionnaire bandwidth. Analysis of items administered and correlations will indicate on unsuitable and congruent items which will be removed from research. In the second part of the study 100 female participants will be nominated for research. Participants will be briefed about the research rationale and procedure and instructed to sign an informed consent (parents of minors will be briefed and instructed to sign as well) indicating on their willingness to participate. Following this participants will be administered interviews, self report questionnaires and computerized tasks by the research team. It will be clarified to participants that questionnaires are anonymous and there are no wrong or right answers. Participants that are not able to handle research demands due to their physical condition will be interviewed by the research team in accordance with the nature of the questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Psychiatric Diagnosis of Bulimia Nervosa, Anorexia Nervosa

Exclusion Criteria:

* BMI < 16

Ages: 13 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: For our research we will recruit 100 participants from a sample of female patients, diagnosed with Eating Disorders and suicidal behavior, admitted to mental health departments in general and psychiatric hospitals. Diagnosis will be made by the hospital staff. After receiving approval from the medical staff participants will be interviewed, handed questionnaires and computerized tasks.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
impulsive tendency | throughout study completion, approximately 1 year
  computerized tasks

SECONDARY OUTCOMES:
impulsivity self report | throughout study completion, approximately 1 year
  questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Yari Gvion, DR, Study Director — Bar Ilan University